CLINICAL TRIAL: NCT05502978
Title: Effect of Education Using WhatsApp and Face-to-Face Meetings Concerning Infant and Young Child Feeding in the COVID-19 Pandemic on the Nutritional Status of Infants: Protocol for a Prospective Interventional Study
Brief Title: Education Using WhatsApp and Face-to-Face Meetings on IYCF for the Nutritional Status of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Eka Nurhayati, Principal investigator, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 110289
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Nutritional Stunting
Keywords: blended education; Infant and Young Child Feeding; Nutritional status of Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The intervention group is third trimester pregnant women with 37 weeks of gestation who received blended education. Blended education is provided by cadres and nutritionists, both online and offline. Education consists of online assistance with digital booklets, videos via WhatsApp by cadres and consultation with nutritionists as well as home visits (offline/face-to-face) by cadres and the research team. One education is done during the third trimester at 37 weeks of gestation, second education is done at 38 weeks' gestation, the third education is done when the baby is 3 months old, all three of which are done online. Mother will be visited every month by cadres and the research team from birth to 7 month old. Consultation with a nutritionist is carried out via WhatsApp calls at critical times the failure rate in IYCF practice was for infants aged 1 month, 3 months, 6 and 7 months
  Interventions: Behavioral: Blended education of Infant and Young Child Feeding

INTERVENTIONS:
Behavioral: Blended education of Infant and Young Child Feeding — Blended education is an intervention about IYCF consisting of 3 components: Education via WhatsApp group, counselling face to face, Consultation with nutritionist via WhatsApp call. In the intervention group, participants will get blended education about IYCF provided by trained cadres. Education via WhatsApp group. The implementation of this educational program was carried out for 3 meeting sessions, where previously trained cadres had distributed videos and digital booklets for IYCF material and opened a discussion session at the end of the meeting in WhatsApp group. Face to face Counselling (Home visit). The cadres conduct home visits every month when the participants have given birth until the child is 7 months old. Consultation with nutritionist via WhatsApp call. Consultations were carried out via WhatsApp calls about IYCF practice was for infants aged 1 month, 3 months, 6 and 7 months.

SUMMARY:
The COVID-19 pandemic affects all activities, including stunting prevention. Almost all cities implement Internet-based learning can be used as an alternative to providing education and allows to exchange personal experiences and also establish interpersonal relationships. Education is one of the intervention efforts that aims to foster and improve the health status of the community, while counselling is a technical part of the educational process itself. blended counselling is the integration of online and offline counselling. Blended counselling is a strategy in the covid-19 pandemic condition and after pandemic. the virtual Education method has also been widely used around the world. The WhatsApp application ranks 2 among the most popular social media in Indonesia.

Blended education innovations are offered online in the form of digital booklets, videos, online discussions, and online consultations carried out via WhatsApp and offline visits according to health protocols. This blended education is expected to facilitate the work of cadres in providing Infant and young child feeding (IYCF) education, to improve IYCF practices for infant nutritional status.

DETAILED DESCRIPTION:
The selection of the research group as the intervention and control group was done by random allocation. Respondents were recruited by self-selection conducted by the research team and the sampling method within the group (treatment group and control group) used was purposive sampling. Recruitment was carried out by means of respondent data obtained from community health center data. Mothers who met the criteria were then included as the research sample. The sample size in this study was determined based on the formula for hypothesis testing on the following two population averages (Lemeshow, et al, 1997). the minimum sample size for the intervention and control groups from previous studies (saleem, et al, 2014) with the results of each group the number of participants for each group of 57 participants plus 10% lost to follow-up, which is 6. the minimum number of samples is 63 samples so that the total number of a minimum sample of 126 respondents.

Participants were recruited by self-selection conducted by the research team and the sampling method within the group (intervention group and control group) used was purposive sampling. Recruitment was carried out by means of respondent data obtained from Primary health care data. Mothers who meet the criteria are then included as research samples. All eligible pregnant women who refer to primary health care for prenatal care at 36-40 weeks of gestation will be requested to participate in the study.

The study uses quantitative data collection methods to evaluate the process and outcome of blended education program. The IYCF assessment include questions regarding demographic data, including age, education, employment status, social economic status, and birth spacing for descriptive information.

The question pre-test post-test for cadres and IYCF education and counselling practice were drawn from IYCF counselling module ministry of health 2014. To assessed the quality of the trainers (research team, nutrition workers for IYCF counsellors and lactation counsellors), clarity of IYCF materials, presentations and training locations were drawn from the questionnaire developed by the researcher. The result effect education for participants by cadre assess using the questionnaire knowledge breastfeeding, responsive feeding and complementary feeding, attitude breastfeeding, self-efficacy breastfeeding and complementary-feeding. the validity and reliability of the questionnaire were tested.

The question pre-test post-test for participants using the questionnaire knowledge breastfeeding, responsive feeding and complementary feeding, attitude breastfeeding, self-efficacy breastfeeding and complementary-feeding. the validity and reliability of the questionnaire were tested. To assessed the quality of the cadre clarity of IYCF materials, presentations and WhatsApp media education were drawn from the questionnaire developed by the researcher. the research team and cadre will assess the respondent (using a questionnaire) about IYCF practice. The data taken at the time of observation were early initiation of breastfeeding, exclusive breastfeeding, breastfeeding >6 months, complementary feeding and continued breastfeeding. Anthropometric measurements for infant nutritional status were carried out from birth to 7 months of age. Bodyweight, height, and head circumference were measured by cadres accompanied by research assistants. Measurement of weight and height using GAMAKIDS, while head circumference using a tape measure. Measurements were taken once a month at the same time, without wearing clothes.

Plan for missing data will be used regression imputation and last observation carried forward. In regression imputation, the existing variables are used to make a prediction, and then the predicted value is substituted as if an actual obtained value. This studies are performed with the longitudinal or time-series approach, in which the subjects are repeatedly measured over a series of time-points because the blended education intervention start from birth to 7 month old. This method replaces every missing value with the last observed value from the same subject. Whenever a value is missing, it is replaced with the last observed value.

Descriptive statistics will be used for baseline data. the collected data will be analyzed in the SPSS software (version 20) using descriptive statistics, such as frequency distribution tables. Also, T-test to see the difference in the average scores between the intervention group and the control group, as well as the pretest-posttest value, namely the influence of the blended education from antenatal period about IYCF on maternal knowledge, attitudes, and self-efficacy. A Chi-square test was also carried out to determine the relationship between two variables whose measurement parameters have been categorized.

One-way analysis of variance (ANOVA) will be used to the effect of blended education from antenatal period about IYCF on infant nutritional status together with knowledge, attitude, self-efficacy, and infection status. The confounding factors and the effect of modifier, stratification analysis was used mantel hanzel's test. The p value of less than 0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are currently pregnant for the first or second time
* Mother does not have chronic disease such as asthma, hypertension and coronary heart disease
* Planning to stay minimal for a year in the research area
* Having smartphone with access to internet and whatsApp messaging application

Exclusion Criteria:

* Participants who have multiple pregnancies
* After the baby was born has a congenital disease/congenital disorders
* Participants unwilling to continue with the study

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Infant Nutritional status | birth to 7 months
  The baby's body condition is determined by the TB/U indicator (according to the WHO-MGRS standard book), nominal scale, body lenght measurement using Infantometer,1=stunting if TB/U <-2 SD 2= not stunting if TB/U -2 SD to < 3 SD, The higher scores mean a better nutritional status of infant
Infant and young child feeding practice (early initiation of breastfeeding practice) | at birth to one hour
  The process of breastfeeding that begins as soon as possible, immediately after birth by allowing the baby to make skin-to-skin contact with the mother's skin for at least the first hour after birth, nominal scale, Measurement using a questionnaire
Infant and young child feeding practice (Exclusive breastfeeding practice) | at birth to 6 months
  The mother's behaviour is to give only breast milk without any additional food/drink, except for drugs or vitamins from birth to 6 months of age. nominal scale. Measurement using a questionnaire
Infant and young child feeding practice (complementary feeding practice) | 6 months to 7 months
  Complementary feeding activities are carried out by providing food at the right time and adequate in terms of quantity, ratio scale, measurement using a questionnaire,The higher scores mean a better practice complementary feeding.
Infant and young child feeding practice (continued breastfeeding >6 month practice) | 6 months to 7 months
  Breastfeeding at the age of > 6 months as an additional consumption of complementary foods for breast milk, ordinal scale, measurement using a questionnaire, not good=given <10 times, good=given >10 times,The higher scores mean a better practice

SECONDARY OUTCOMES:
Changes in knowledge breastfeeding | 37 weeks gestation to the child is 4 months
  Ability to give precise answers to questions regarding breastfeeding, interval scale,measurement using a questionnaire totaling 15 items. The value is Poor knowledge (0-10), enough knowledge (11-20), Good knowledge (21-30). The higher scores mean a better knowledge about breastfeeding
Changes in attitude breastfeeding | 37 weeks gestation to the child is 6 months
  Responses to breastfeeding in the cognitive, affective and psychomotor domains. All items are measured using a 4-point Likert scale, interval scale, measurement using a questionnaire
Changes in self-efficacy breastfeeding | 37 weeks gestation to the child is 6 months
  Self-efficacy breastfeeding measurement is the score obtained by the research subjects through the responses given to the Breastfeeding Self Efficacy Scale Short Form (BSES-SF) scale, BSES consist of 14 items, ordinal scale, measurement using a questionnaire,The higher score of the the self-efficacy, the better the respondent's self-efficacy
Changes in knowledge complementary feeding | 37 weeks gestation to the child is 7 months
  Ability to give correct answers to questions regarding complementary feeding, interval scale,measurement using a questionnaire totaling 20 items. The value is Poor knowledge (0-13), enough knowledge (14-27), Good knowledge (28-49). The higher scores mean a better knowledge about complementary feeding.
Changes in self-efficacy complementary feeding | 37 weeks gestation to the child is 7 months
  Self-efficacy complementary feeding is mother's belief and confidence to carry out complementary feeding activities by providing food at the right and adequate time. ratio scale, measurement using a questionnaire,The higher score of the self-efficacy, the better the respondent's self-efficacy
Changes in knowledge of cadre | one week
  Knowledge measurement is ability to provide precise answers to questions regarding about infant and young child feeding,Interval scale, measurement using a questionnaire totalling 15 items.The value is Poor knowledge (1-5), enough knowledge (6-10), Good knowledge (11-15). The higher scores mean a better knowledge of cadres.
Changes in practice counselling of cadre | 37 weeks gestation to the child is 7 months
  Practice is the ability of cadres to provide counselling to participants, interval scale, measurement using a questionnaire totalling 26 items. The value is poor practice (0-8), enough practice (9-17), good practice (18-26). The higher scores mean a better practice counselling of cadres.

CONTACTS AND LOCATIONS:
Overall Officials: Siti Helmyati, ph.D, Study Director — Gadjah Mada University
Locations (3):
- Indonesia (3):
  - Sewon community health center, Bantul, Special Region of Yogyakarta
  - Pandak community health center, Bantul, Special Region of Yogyakarta
  - Bambanglipuro Health centre, Bantul, Special Region of Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Epstein A, Moucheraud C, Sarma H, Rahman M, Tariqujjaman M, Ahmed T, Glenn J, Bossert T, Kruk ME. Does health worker performance affect clients' health behaviors? A multilevel analysis from Bangladesh. BMC Health Serv Res. 2019 Jul 24;19(1):516. doi: 10.1186/s12913-019-4205-z. PMID 31340809
- [Result] Mousavi SR, Amiri-Farahani L, Hasanpoor-Azghady SB, Saravi SO. Comparing the effect of in-person and virtual childbirth preparation trainings on the fear of childbirth (FOC) and pregnancy experience of pregnant women: protocol for a quasi-experimental feasibility study. Pilot Feasibility Stud. 2021 Nov 5;7(1):194. doi: 10.1186/s40814-021-00933-w. PMID 34740371
- [Result] Susiloretni KA, Hadi H, Prabandari YS, Soenarto YS, Wilopo SA. What works to improve duration of exclusive breastfeeding: lessons from the exclusive breastfeeding promotion program in rural Indonesia. Matern Child Health J. 2015 Jul;19(7):1515-25. doi: 10.1007/s10995-014-1656-z. PMID 25487415
- [Result] Susiloretni KA, Hadi H, Blakstad MM, Smith ER, Shankar AH. Does exclusive breastfeeding relate to the longer duration of breastfeeding? A prospective cohort study. Midwifery. 2019 Feb;69:163-171. doi: 10.1016/j.midw.2018.11.008. Epub 2018 Nov 19. PMID 30522038
- [Result] Kang H. The prevention and handling of the missing data. Korean J Anesthesiol. 2013 May;64(5):402-6. doi: 10.4097/kjae.2013.64.5.402. Epub 2013 May 24. PMID 23741561
- [Result] Saleem AF, Mahmud S, Baig-Ansari N, Zaidi AK. Impact of maternal education about complementary feeding on their infants' nutritional outcomes in low- and middle-income households: a community-based randomized interventional study in Karachi, Pakistan. J Health Popul Nutr. 2014 Dec;32(4):623-33. PMID 25895196
- [Result] Hosmer DW, Hosmer T, Le Cessie S, Lemeshow S. A comparison of goodness-of-fit tests for the logistic regression model. Stat Med. 1997 May 15;16(9):965-80. doi: 10.1002/(sici)1097-0258(19970515)16:93.0.co;2-o. PMID 9160492
- See also: Blended counselling a means of supporting students University of Eastern Finland — http://www.oppi.uef.fi/wanda/virtukampus/wp-
- See also: UNICEF/WHO/World Bank Group Joint Child Malnutrition Estimates — http://data.unicef.org/wp-content/uploads/2018/05/JME-2018-brochure-web.pdf.